CLINICAL TRIAL: NCT04699318
Title: To Compare the Frequency of Urethrocutaneous Fistula After Double Dartos Tubularized Incised Plate (TIP) Urethroplasty and Single Dartos Tubularized Incised
Brief Title: Urethrocutaneous Fistula Rate After Double Dartos and Single Dartos Tubularized Incised Plate Urethroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Malik Asad Munir, Malik ASAD Munir, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEMU1234
Record Dates: First submitted 2018-11-05; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Dartos TIP (Experimental): Single dartos tubularized incised plate urethroplasty
  Interventions: Procedure: Group A
- Double Dartos TIP (Experimental): Double dartos tubularized incised plate urethroplasty
  Interventions: Procedure: Group B

INTERVENTIONS:
Procedure: Group B — To release the pediatric hypospadias using Double Dartos Tubularized incised plate (TIP) Urethroplasty
  Other Names: Double dartos TIP
  Arms: Double Dartos TIP
Procedure: Group A — To release the pediatric hypospadias using Single Dartos Tubularized incised plate (TIP) Urethroplasty
  Other Names: Single dartos TIP
  Arms: Single Dartos TIP

SUMMARY:
The subjects were divided into two groups. Each group comprised 30 children. Children were randomly allocated in two groups via computer generated tables. Children in group-A underwent single dartos tubularized incised plate urethroplasty while those in group-B underwent double dartos tubularized incised plate urethroplasty.

DETAILED DESCRIPTION:
In group A dartos flap is raised from foreskin of the patient and applied as a single layer after tubularization in between neourethra and skin . In group B dartos flap is raised from the foreskin of patient and divided in two equal halves.Both flaps are placed as two layers in between skin and neourethra.After surgery patient is kept in ward for 10 days with stent.Patient is followed up in OPD on after 7th day after discharge for outcome.

ELIGIBILITY:
Inclusion Criteria All the patients above one year of age All patients having distal and mid penile hypospadias. -

Exclusion Criteria Severe chordee Previously operated cases Patient with undescended testis Circumcised patient

-

Ages: 2 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male gender
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Recurrence of urethro-cutaneous fistula | 17 days
  Abnormal communication between urethra and penile skin after urethroplasty, presenting with complaints of two streams of micturition and noted on examination at 17th postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Asad Munir, FCPS, Principal Investigator — King Edward Medical University
Locations (1):
- KEMU, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided